CLINICAL TRIAL: NCT00296985
Title: The Impact of Continuous Flow Cellsaver on Neurocognitive Decline After Cardiac Surgery
Brief Title: Continuous Cellsaver and Neurocognitive Decline Post Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UHN REB 01-0420-B; HSFO NA4915
Record Dates: First submitted 2006-02-23; First posted 2006-02-27 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Heart Disease; Neurocognitive Decline
Keywords: Cardiac surgery; Cellsaver; Neurocognitive Function; Neuronal Protection; Quality of Life
MeSH Terms: conditions — Heart Diseases

INTERVENTIONS:
Device: Fresenius Cellsaver

SUMMARY:
Patients having cardiac surgery to correct their heart disease may suffer a decline in mental and neurologic abilities. Passage of small particles of fat, tissue waste and air bubbles to the brain while on the heart-lung machine is thought to be one cause for decline in mental and neurologic abilities (the function of brain) after surgery.

The purpose of this study is to determine if replacement of cardiotomy suction (one part of the heart-lung machine) with the cell-saver (a different part of the heart-lung machine) during surgery will help to prevent a decline in mental and neurologic abilities after surgery. investigating 312 patients over 2 years,patients will be assigned randomly to either cardiotomy suction or cell-saver group. Patients will be given questionnaires before surgery, 6 weeks and 1-year after surgery. These questionnaires will assess memory, attention span, the ability to concentrate and the quality of life. Patients will also have a brief neurologic exam (physical examination to check mental state, reflexes, strength, and balance) before surgery, 3-5 days after surgery, 6 weeks and 1-year after surgery to determine any changes. Cell-saver separates red blood cells from tissue waste products and fat prior to returning blood back to the patient and may reduce the negative effects of particles of fat, tissue waste and air bubbles have on the brain. Potential benefits of cell-saver device when used during surgery may prevent the decrease in memory, attention span, and the ability to concentrate resulting in improved quality of life after surgery.

Objectives: The primary aim is to determine the effect of continuous flow cell-saver on short and long term neurocognitive function after cardiac surgery, measured by precise preoperative and postoperative psychometric and neurologic testing. Hypothesis: The primary hypothesis: Continuous flow cell-saver reduces postoperative neurocognitive decline following cardiac surgery. Methodology: 312 informed and consenting patients, age > 65 years, scheduled for coronary artery bypass graft surgery will be prospectively enrolled over a 2-year period. Patients will be randomly allocated to either the continuous flow cell-saver or conventional cardiotomy suction (controls). Neurological history and physical exam will be completed preoperatively, discharge, 6-weeks and 1-year after surgery. Transcranial Doppler scanning will be used for intraoperative monitoring of cerebral embolic load. Transesophageal echocardiography and epiaortic scanning will be employed to account for the severity of the aortic atheroma scores. Neurocognitive testing and quality of life assessment will be conducted preoperatively , 6-weeks and 1-year after surgery. Significance: The utilization of continuous flow cell-saver may reduce the negative effects of fat particles, tissue waste and air emboli have on brain.

ELIGIBILITY:
Inclusion Criteria:

* Age > 65 years,
* elective CABG surgery
* signed informed consent

Exclusion Criteria:

* Severe kidney (creatinine > 2.5mg/dL and
* liver disease (bilirubin > 2 mg/dL)
* symptomatic cerebrovascular disease
* alcoholism
* psychiatric illness
* patients who are unable to read or who have less than a 7th grade education.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312
Dates: Start 2001-12; Primary Completion 2005-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
The primary aim is to determine the effect of continuous flow cell-saver on short and long term neurocognitive function after cardiac surgery, measured by preoperative and postoperative psychometric and neurologic testing. | 1 year

SECONDARY OUTCOMES:
A secondary aim is to determine if the improvement in cognitive function is associated with improved quality of life after cardiac surgery. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: George N Djaiani, MD, Principal Investigator — Toronto General Hospital, University Health Network
Locations (1):
- Toronto General Hospital, University Health Network, Toronto, Ontario, Canada